CLINICAL TRIAL: NCT06032702
Title: Effect of 3 Week vs 6 Week Orthodontic Appointment Intervals on Teeth Alignment in Patients With Moderate to Severe Dental Crowding: a Randomized Clinical Trial
Brief Title: Effect of 3 Week vs 6 Week Orthodontic Appointment Intervals on Teeth Alignment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bkahtawar Amin Medical and Dental College Multan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAMDC 0001
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Orthodontic Tooth Movement; Tooth Alignment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 week interval (Experimental): 3 week orthodontic interappointment interval
  Interventions: Procedure: tooth alignment
- 6 week interval (Experimental): 6 week orthodontic interappointment interval
  Interventions: Procedure: tooth alignment

INTERVENTIONS:
Procedure: tooth alignment — Alignment will be assessed by Little's Irregularity Index

SUMMARY:
Effect of 3 week vs 6 week orthodontic appointment intervals on teeth alignment in patients with moderate to severe dental crowding: a randomized clinical trial.

There is still inconclusive evidence about the orthodontics treatment duration and interappointment interval.

DETAILED DESCRIPTION:
Patients with moderate to severe crowding will be divided randomly into two groups (Group A and Group B). Group A includes patients with an interval of 3 weeks between their appointments while Group B includes the patients with an interval of 6 weeks between their appointments.

1. To determine the mean changes in the tooth irregularity index of a patient with mild to moderate crowding activated every 3rd week
2. To determine the mean changes in the tooth irregularity index of a patient with mild to moderate crowding activated every 6th week
3. To compare the difference between the two modalities in percentage

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16-30
* Little's irregularity index from 5mm to 12mm
* Healthy periodontium
* No systemic disease
* Patients giving consent for inclusion

Exclusion Criteria:

* Little's irregularity index less than 5mm and more than 12mm
* Blocked out incisors needing push coil
* Ankylosed teeth
* Active periodontal disease
* Systemic bone disease
* Non-compliant patients
* Patients with frequent breakages

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
alignment efficiency and interappointment interval | Time frame for measurement of (Little's Irregularity Index) was every 6th week over a period of 6 months, giving a total of 5 measurements
  Changes in Little's Irregularity Index between arm 1 and arm 2 and comparison of both interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakhtawar Amin Medical And Dental College, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Undecided